CLINICAL TRIAL: NCT00835107
Title: An Investigation of Sleep Architecture in Ziprasidone-Treated Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Providence Health & Services (Other); Pfizer (Industry); MDS Pharma Services (Industry)
Responsible Party: Principal Investigator, Dr. Roumen Milev, MD, PhD, FRCPsych, FRCPC, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSIY-287-08; GA128250
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Depression, Bipolar
Keywords: Bipolar Depression; Sleep; Polysomnograph; Slow Wave Sleep; Ziprasidone; Antipsychotic; Placebo
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ziprasidone (Experimental)
  Interventions: Drug: ziprasidone hydrochloride
- Sugar pill (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ziprasidone hydrochloride — oral capsules, from 40-80 mg BID, for one month with the option to continue the medication after the study has been completed
  Other Names: Zeldox
  Arms: Ziprasidone
Drug: placebo — placebo comparator, oral capsules, BID, for one month
  Arms: Sugar pill

SUMMARY:
This study uses polysomnographs(PSG) to investigate sleep patterns in patients with bipolar depression. This is a double-blind, placebo-controlled, study of ziprasidone that is added to patients current medications. The objective is to relate changes in slow wave and rapid eye movement sleep to changes in mood and overall illness severity. Participants will be randomly assigned to add either placebo or ziprasidone to their current treatment regimen. Participants make 3 to 4 study visits, over a 1 month period, at which they will be asked about their history, mood and sleep quality. Participants will also have three in-home overnight polysomnographs.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Bipolar Disorder Type 1,2 or NOS by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV).
* Current depressive episode with a HAMD-17 of >16.
* Males or Females over age 18yrs.
* Inpatients or outpatients.
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment.
* Able to understand and comply with the requirements of the study.
* Provision of written informed consent.

Exclusion Criteria:

* Current Manic, Hypomanic or Mixed episode, with YMRS > 12.
* Current or past diagnosis of Schizophrenia and Dementia.
* Pregnant women, or women in childbearing age, not willing to use appropriate contraception or women currently nursing.
* Patient on any other antipsychotic medication.
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others.
* Known intolerance or lack of response to Ziprasidone, as judged by the investigator.
* Benzodiazepines and all other sleep-aids must be discontinued prior to participation in the study if they have not been at a stable dosage for the 4 weeks previous to entry into the study.
* No change to the current medication regime (excluding discontinuation of sleep aids and antipsychotic medications) is allowed 4 weeks prior to the first PSG reading.
* Administration of a depot antipsychotic injection within two dosing interval (for the depot) before randomization.
* Substance or alcohol dependence at enrolment or in the last three months (except for caffeine or nicotine dependence), as defined by DSM-IV criteria.
* Serious, unstable or inadequately treated medical illness as judged by the investigator.
* History of epilepsy or uncontrolled seizures.
* Involvement in the planning and conduct of the study.
* Previous enrolment in the present study.
* Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements.
* Patients with serum potassium, magnesium and/or calcium levels outside the normal range at baseline.
* Patients with marked liver function abnormalities at baseline, demonstrated by laboratory values, by judgment of the investigator.
* Known serological evidence of HIV, or acute or chronic hepatitis; donation of blood or blood products for transfusion prior to initiation of the treatment with study drug, during the study and for 30 days after the study has ended.
* Known history of QT prolongation (including congenital long QT syndrome).
* Recent acute myocardial infarction or uncompensated heart failure.
* Currently taking other drugs that are known to prolong the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To assess the objective (polysomnographic) changes in sleep quality before and after introduction of Ziprasidone in treatment of patients with bipolar depression. | 1 month

SECONDARY OUTCOMES:
To assess the subjective changes in sleep quality parameters before and at different stages after introduction of ziprasidone in treatment, longitudinally, and to correlate these changes with measures of illness severity. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Roumen Milev, MD, Principal Investigator — Queen's University; Anusha Baskaran, BScH, Principal Investigator — Queen's University
Locations (1):
- Providence Care Mental Health Services, Kingston, Ontario, Canada

REFERENCES:
- [Background] Cohrs S, Meier A, Neumann AC, Jordan W, Ruther E, Rodenbeck A. Improved sleep continuity and increased slow wave sleep and REM latency during ziprasidone treatment: a randomized, controlled, crossover trial of 12 healthy male subjects. J Clin Psychiatry. 2005 Aug;66(8):989-96. doi: 10.4088/jcp.v66n0805. PMID 16086613
- [Background] Sharpley AL, Cowen PJ. Effect of pharmacologic treatments on the sleep of depressed patients. Biol Psychiatry. 1995 Jan 15;37(2):85-98. doi: 10.1016/0006-3223(94)00135-P. PMID 7718684